CLINICAL TRIAL: NCT02999373
Title: Autologous Cord Blood Mononuclear Cells for Bronchopulmonary Dysplasia in Very Preterm Neonates
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, yang jie, Professor, Guangdong Women and Children Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Guangdong M And C
Record Dates: First submitted 2016-12-03; First posted 2016-12-21 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Bronchopulmonary Dysplasia; Premature; Neonatal Death
Keywords: prevention; Bronchopulmonary Dysplasia; preterm; cord blood mononuclear cells
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth; Perinatal Death

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous cord blood mononuclear cells (Experimental): Autologous Umbilical Cord Blood Mononuclear Cells Therapy 24 hours after birth ,dose is 50 million cells/kg
  Interventions: Other: Autologous Umbilical Cord Blood Mononuclear Cells Therapy
- control (No Intervention)

INTERVENTIONS:
Other: Autologous Umbilical Cord Blood Mononuclear Cells Therapy — Autologous Umbilical Cord Blood Mononuclear Cells Therapy in preterm for prevention of infection
  Arms: Autologous cord blood mononuclear cells

SUMMARY:
Rationale: Pre-clinical animal studies provide robust evidence regarding the beneficial effect of cord blood-derived mononuclear cells (MNCs) for experimental bronchopulmonary dysplasia (BPD).

This single-center, non-randomized, controlled, blinded trial assessed the effect of a single intravenous infusion of autologous cord blood MNCs (ACBMNCs) in preventing BPD in very preterm neonates, a high-risk population.

ELIGIBILITY:
Inclusion Criteria: (1) born at the study hospital; (2) singleton birth; (3) GA <32 weeks; (4) free of severe congenital anomalies or genetic syndromes; (5) without clinical chorioamnionitis; (6) the mother was negative for hepatitis B (HBsAg and/or HBeAg), hepatitis C (anti-HCV), syphilis, HIV (anti-HIV-1 and -2), and IgM against cytomegalovirus, rubella, toxoplasma, and herpes simplex viruses; (7) consent was obtained from the parents or guardians; and (8) after processing, UCB cells were available.

Ages: 0 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
bronchopulmonary dysplasia at 36 weeks of postmenstrual age or the discharge home | 36 weeks of postmenstrual age or the discharge
  bronchopulmonary dysplasia rate

SECONDARY OUTCOMES:
number of patients with severe BPD in survivors | 36 weeks of postmenstrual age or the discharge
  severe BPD in survivors
number of patients died before discharge from hospital | before discharge from hospital
  mortality before discharge from hospital
the duration of mechanical ventilation | before discharge from hospital
  Other outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yang, PHD, Principal Investigator — Guangdong Women and Children Hospital
Locations (1):
- Jie Yang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ballen KK, Gluckman E, Broxmeyer HE. Umbilical cord blood transplantation: the first 25 years and beyond. Blood. 2013 Jul 25;122(4):491-8. doi: 10.1182/blood-2013-02-453175. Epub 2013 May 14. PMID 23673863
- [Background] Mezey E, Nemeth K. Mesenchymal stem cells and infectious diseases: Smarter than drugs. Immunol Lett. 2015 Dec;168(2):208-14. doi: 10.1016/j.imlet.2015.05.020. Epub 2015 Jun 4. PMID 26051681
- [Background] Wannemuehler TJ, Manukyan MC, Brewster BD, Rouch J, Poynter JA, Wang Y, Meldrum DR. Advances in mesenchymal stem cell research in sepsis. J Surg Res. 2012 Mar;173(1):113-26. doi: 10.1016/j.jss.2011.09.053. Epub 2011 Oct 24. PMID 22225756
- [Background] Leung, Kam Tong; Lam, Hugh Simon; Chan, Kathy Yuen Yee, Decreased Frequency of Circulating CD34+Hematopoietic Stem/Progenitor Cells in Preterm Infants with Late-Onset Systemic Bacterial Infection,Blood,2014.124.21
- [Background] Lam HS, Cheung HM, Poon TC, Wong RP, Leung KT, Li K, Ng PC. Neutrophil CD64 for daily surveillance of systemic infection and necrotizing enterocolitis in preterm infants. Clin Chem. 2013 Dec;59(12):1753-60. doi: 10.1373/clinchem.2013.209536. Epub 2013 Sep 17. PMID 24046202
- [Background] Ho MS, Mei SH, Stewart DJ. The Immunomodulatory and Therapeutic Effects of Mesenchymal Stromal Cells for Acute Lung Injury and Sepsis. J Cell Physiol. 2015 Nov;230(11):2606-17. doi: 10.1002/jcp.25028. PMID 25913273
- [Background] van den Berg JP, van Zwieteren N, Westerbeek EA, Garssen J, van Elburg RM. Neonatal modulation of serum cytokine profiles by a specific mixture of anti-inflammatory neutral and acidic oligosaccharides in preterm infants. Cytokine. 2013 Oct;64(1):188-95. doi: 10.1016/j.cyto.2013.07.002. Epub 2013 Aug 2. PMID 23911205
- [Background] Lam HS, Wong SP, Liu FY, Wong HL, Fok TF, Ng PC. Attitudes toward neonatal intensive care treatment of preterm infants with a high risk of developing long-term disabilities. Pediatrics. 2009 Jun;123(6):1501-8. doi: 10.1542/peds.2008-2061. PMID 19482760
- [Background] Strunk T, Inder T, Wang X, Burgner D, Mallard C, Levy O. Infection-induced inflammation and cerebral injury in preterm infants. Lancet Infect Dis. 2014 Aug;14(8):751-762. doi: 10.1016/S1473-3099(14)70710-8. Epub 2014 May 28. PMID 24877996
- [Derived] Ren Z, Yang L, Wang J, Han J, Lin S, Yao Y, Du C, Yang J. Cord blood stem cell-derived Angptl7 ameliorates the severity of bronchopulmonary dysplasia via anti-inflammatory and proangiogenic effects. Mol Med Rep. 2024 Jan;29(1):8. doi: 10.3892/mmr.2023.13131. Epub 2023 Nov 24. PMID 37997800
- [Derived] Zhuxiao R, Fang X, Wei W, Shumei Y, Jianlan W, Qiuping L, Jingjun P, Chuan N, Yongsheng L, Zhichun F, Jie Y. Prevention for moderate or severe BPD with intravenous infusion of autologous cord blood mononuclear cells in very preterm infants-a prospective non-randomized placebo-controlled trial and two-year follow up outcomes. EClinicalMedicine. 2023 Feb 16;57:101844. doi: 10.1016/j.eclinm.2023.101844. eCollection 2023 Mar. PMID 36864985